CLINICAL TRIAL: NCT00424086
Title: Single Blind, Randomized, Actively Controlled Phase 1/2 Study to Compare the Safety and Immunogenicity of a Split Virus, Vero Cell Derived, Seasonal Influenza Vaccine (VCIC) With a Licensed, Egg Derived, Split Virus, Seasonal Influenza Vaccine (EIV)
Brief Title: Safety and Immunogenicity Study of an Inactivated Influenza Vaccine (Split Virus, Vero Cell Derived)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 720601
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2008-01

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Inactivated seasonal influenza vaccine (split virus, vero cell derived)
Biological: Inactivated seasonal influenza vaccine (split virus, egg derived) [licensed control vaccine]

SUMMARY:
The objective of this study is to assess the safety, tolerability and immunogenicity of a Split Virus, Vero Cell derived, Seasonal Influenza Vaccine (VCIV) in comparison to a Licensed Egg Derived, Split Virus, Seasonal Influenza Vaccine (EIV) in healthy subjects 18 years of age and older.

Approximately 1000 subjects will be randomly assigned in a 3:1 ratio to receive a single injection of VCIV or EIV. Subjects will be monitored for 180 days following vaccination for occurrence of adverse reactions and for antibody response to the vaccine.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects who

* Are 18 to 49 years of age (inclusive) on the day of screening (Stratum A)
* Are 50 years of age or older on the day of screening (Stratum B)
* Have an understanding of the study, agree to its provisions, and give written informed consent prior to study entry
* Are clinically healthy (in a physical condition such that the physician would have no reservations administering influenza vaccine outside the scope of a clinical study)
* Are physically and mentally capable of participating in the study
* Agree to keep a daily record of symptoms
* If female and capable of bearing children, have a negative urine pregnancy test result within 24 hours of the vaccination on Study Day 0 and agree to employ adequate birth control measures. For the purposes of this study adequate birth control measures incorporate 2 types of the following FDA approved birth control measures through 60 days after vaccination:

  * Hormonal types of birth control (such as implants, birth control pills, patches or other methods) or an intrauterine device, AND
  * An additional barrier type of birth control measure (i.e., condoms, diaphragms, cervical caps, etc.)

Exclusion Criteria:

Subjects who

* Have previously been vaccinated against influenza with vaccine formulated for the 2006/2007 influenza season
* Have an oral temperature >=37.5°C at the time of vaccination on Day 0 (see note below)
* Have Type I diabetes
* Have a Body Mass Index >35
* Have hypertension at screening (with or without medication) that is graded as greater than Stage 1 defined as a systolic pressure >159 or diastolic pressure >99 while seated and at rest (measurement may be repeated twice before subject is absolutely excluded)
* Have clinically significant abnormal clinical laboratory values at screening
* Have clinically significant electrocardiographic abnormalities at screening
* Test positive for Human Immunodeficiency Virus(HIV), Hepatitis B Surface Antigen (HbsAg) or Hepatitis C Virus (HCV)
* Have a history of cardiovascular disease that required hospitalization
* Have a history of immunodeficiency or autoimmune diseases
* Have a history of arthritis (joint swelling, tenderness, warmth or erythema) on more than one occasion, not related to trauma (including running) or any episode of non-trauma related arthritis within the previous 6 months
* Suffer from active neoplastic disease or have a history of hematologic malignancy
* Suffer from a disease or are undergoing a form of treatment that can be expected to influence immune response. Such treatment includes, but is not limited to systemic or high dose inhaled (>800 μg/day of beclomethasone dipropionate or equivalent) corticosteroids, radiation treatment or other immunosuppressive or cytotoxic drugs
* Have a history of inflammatory or degenerative neurological disease (e.g. Guillain Barré, multiple sclerosis)
* Have received any vaccination within 2 weeks prior to vaccination in this study
* Have received a blood transfusion or immunoglobulins within 30 days prior to vaccination in this study
* Have donated blood or plasma within 30 days prior to vaccination in this study
* Have a history of any vaccine related contraindicating event (e.g., anaphylaxis, allergy to eggs, allergy to components of the test or comparator vaccine, other known contraindications)
* Have a rash, dermatologic condition or tattoos which may interfere with injection site reaction rating
* Have a positive urine drug screen (unless the detected drug is currently prescribed by a licensed health care provider and the continued administration of the drug would not otherwise exclude the subject from participation)
* Were administered an investigational drug within 6 weeks prior to study entry
* Are concurrently participating in a clinical study that Inactivated Influenza Vaccine (Split Virus, Vero Cell Derived)includes the administration of an investigational product
* Are a member of the team conducting this study
* Are in a dependent relationship with the study investigator. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the investigator
* If female, are pregnant or lactating.

NOTE: If all other inclusion/exclusion criteria are met, a subject with a temperature >=37.5°C on Day 0 may be included in the study at a repeat visit provided:

1. They do not have an oral temperature >=37.5°C at the repeat visit,
2. The repeat visit is no more than 5 calendar days after the initial Day 0 visit,
3. The repeat visit is no more than 21 calendar days after all other screening procedures are completed,
4. Subjects are still being recruited at the study site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2007-01; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of Vero cell derived vaccine in comparison to egg-derived vaccine in healthy subjects in two age strata: 18 to 49 years, and 50 years of age and older
To assess the immunogenicity of Vero cell derived vaccine in comparison to egg-derived vaccine for subjects in two age strata: 18 to 49 years of age and 50 years of age and older

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Investigator, Principal Investigator — Baxter Healthcare Corporation
Locations (8):
- Austria (2):
  - Kinemed, Graz
  - Universitaetsklinik f. Klinische Pharmakologie, Allgemeines Krankenhaus Wien (University Hospital for Clinical Pharmacology, General Hospital of Vienna), Vienna
- Germany (3):
  - MDS Pharma Services Germany GmbH, Hamburg
  - Internistische Gemeinschaftspraxis Dr. Regner & Dr. Schmitt (Group practice for internal medicine), Mainz
  - Harrison Clinical Research, Munich
- Poland (3):
  - Zespol Przychodni Specjalistycznych "DIAB-END-COR" Sp. z o.o., Krakow
  - PANTAMED Sp. z o.o., Olsztyn
  - Niepubliczny Zaklad Opieki Zdrowotnej, Osrodek Zdrowia w Lipsku, Zamość